CLINICAL TRIAL: NCT06089525
Title: Treatment of Complex Pilon Fractures: A Pilot Study Comparing Primary Arthrodesis (PA) to Open Reduction and Internal Fixation (ORIF)
Brief Title: Treatment of Complex Pilon Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Brent Wise, Assistant Professor, University of Kansas Medical Center
Other Study IDs: 00150446
Record Dates: First submitted 2023-09-13; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Pilon Fracture
Keywords: Pilon Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open reduction and internal fixation (ORIF): Patient has underwent ORIF to repair a pilon fracture.
- Primary arthrodesis (PA; ankle fusion): Patient has underwent PA/ankle fusion to repair a pilon fracture.

SUMMARY:
This project intends to compare patient outcomes between patients undergoing ORIF compared to PA, or ankle fusion, following an acute pilon fracture. Limited literature comparing ORIF and ankle fusion as a primary procedure exists. Particularly, no present literature exists examining the novel arthrodesis surgical technique utilized in this study in conjunction with Opal sensor gait analysis data. This study will serve as a pilot study and assess patient gait, degree of pain, functional outcome scores, development of post-traumatic arthritis and/or infection, need for secondary surgery, and return to work time.

ELIGIBILITY:
Inclusion Criteria: Individuals receiving ORIF or PA for a multifragmented acute pilon fracture occuring at the joint surface over the age of 18 from 2018 to present at The University of Kansas Medical Center (KUMC) or Emory University Hospital.

Exclusion Criteria: Anyone under the age of 18 years. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals over the age of 18 that have undergone an ORIF or PA surgery for an acute pilon fracture at either KUMC or Emory University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-12-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Ankle range of motion | Collected only once; from 6 months post-op up to date of death from any cause
  Inversion and eversion range, and flexion versus extension range determined by the use of the Opal sensors
Walking cadence | Collected only once; from 6 months post-op up to date of death from any cause
  Steps per minute as determined by the use of the Opal Sensors
Timed up-and-go | Collected only once; from 6 months post-op up to date of death from any cause
  Time it takes to stand from seated, walk 10 feet forward, turn around, and sit back down, unassisted (determined by the use of the Opal sensors).
Foot and ankle Outcome Score (FAOS) | Collected only once; from 6 months post-op up to date of death from any cause
  Foot and ankle injury patient reported outcome measure (Scores range from 0 to 100, with higher scores indicating better foot and ankle surgical outcomes)
12 Item Short Form Survey (SF-12) | Collected only once; from 6 months post-op up to date of death from any cause
  Patient reported outcome measures regarding health and daily activities (Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning)

SECONDARY OUTCOMES:
Presence of infection and/or post-traumatic arthritis | From the date of surgery up until the date of death from any cause
  Rate of patients being rehospitalized or returning for care beyond what is required due to infection or arthritis
Need for secondary operation | From the date of surgery up until the date of death from any cause
  Number of patients that required follow up surgery to their initially injured ankle
Return to work time | From the date of surgery up until the date of death from any cause
  Number of weeks it took for patients to return to work

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States